CLINICAL TRIAL: NCT02032719
Title: Investigating Improved Self Management in Uncontrolled Systolic Hypertension
Brief Title: Improved Self Management in Uncontrolled Systolic Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Paul Ritvo, Principal Investigator, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-259
Record Dates: First submitted 2014-01-06; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Systolic Hypertension
Keywords: Hypertension, Systolic, Uncontrolled
MeSH Terms: conditions — Isolated Systolic Hypertension; Hypertension; Systolic Murmurs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- smartphone assisted lifestyle coaching (Experimental): 6 months of smartphone assisted lifestyle coaching
  Interventions: Behavioral: smartphone-assisted health coaching
- Lifestyle health coaching (Active Comparator): 6 months of lifestyle health coaching
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: smartphone-assisted health coaching — smartphone with software provides self monitoring of exercise, diet and stress reduction; provision of timely reminders; photo-journaling of meals; secure text messaging
  Arms: smartphone assisted lifestyle coaching
Behavioral: Lifestyle counseling — Lifestyle counseling
  Arms: Lifestyle health coaching

SUMMARY:
Patients who receive smartphone-assisted health coaching will have a significantly lower 24 hour ambulatory blood pressure mean than patients who receive just health coaching

DETAILED DESCRIPTION:
Primary Outcome Measure: Mean 24 hour ambulatory blood pressure

Secondary Outcome Measures: Profile of Mood States-SF Vigor Scale; Satisfaction with Life Scale; Positive and Negative Affect Schedule; Hospital Anxiety and Depression Scale; SF - 12

ELIGIBILITY:
Inclusion Criteria:

* 25 - 70 years old;
* mean daytime systolic BP> 130 mm. Hg.

Exclusion Criteria:

* Severe or end-stage organ disease (liver, kidney, heart, lung) or history of diabetic ketoacidosis, or any other illness with expected survival less than 1 year;
* severe cognitive impairment;
* diagnosed psychiatric illness or disability;
* clinical significant cardiac arrhythmia;
* symptomatic orthostatic hypertension;
* pregnancy;
* not fluent in english.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
24 hour ambulatory blood pressure mean | 6 months follow up from baseline
  24 hour ambulatory blood pressure assessed at baseline and 6 months follow up in experimental and control groups

SECONDARY OUTCOMES:
Quality of life self report measures | Baseline and 6 months followup
  Profile of Mood States - SF Vigor Scale Satisfaction with Life Scale Positive and Negative Affect Schedule Hospital Anxiety and Depression Scale; SF 12

CONTACTS AND LOCATIONS:
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada